CLINICAL TRIAL: NCT05130905
Title: Safety and Efficacy of a Multivitamin, Multimineral, Bovine Colostrum Containing Supplement RiteStart: An Open Label Trial
Brief Title: RiteStart Personal Nutritional Dietary Study
Acronym: RESPOND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 4Life Research, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RSC-012-00
Record Dates: First submitted 2021-10-22; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Healthy Nutrition
Keywords: Immunity; Salivary IgA; Bovine Colostrum; Brain Health; Heart Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supplementation with RiteStart (Experimental): Once enrolled into the study, participants were instructed to take RiteStart Supplement daily for 12 weeks.
  Interventions: Dietary Supplement: RiteStart Supplement

INTERVENTIONS:
Dietary Supplement: RiteStart Supplement — RiteStart is a comprehensive multivitamin, multimineral, all-in-one daily supplement. Besides having comprehensive and balanced amounts of essential vitamins and minerals that the human body needs, RS includes many other health-promoting ingredients. For example, RS contains potent antioxidants, including vitamins A, C, and E, oligomeric proanthocyanidins from pinebark and grapeseed extracts, lutein, CoQ10, alpha-lipoic acid, and green tea. It is also a source of essential fatty acids from fish and plant oils. RS contains transfer factor (bovine colostrum and egg yolk extracts) that support immunity [6, 7, 8]. RS also includes a blend of maitake mushrooms, shiitake mushrooms, cordyceps, inositol hexaphosphate, olive leaf extract, and other ingredients that aim to further support immune function and overall health.

SUMMARY:
This study is undertaken to explore the effects of a bovine colostrum containing MVM (RiteStart) on different health aspects by quantitatively assessing relevant serum and saliva biomarkers, over a 12-week period in participants.

DETAILED DESCRIPTION:
Blood samples were drawn by a certified phlebotomist, prepared, and then analyzed by a Clinical Laboratory Improvement Amendments (CLIA)-certified independent laboratory. The following components were measured in sera from the participants: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Gamma-Glutamyl Transpeptidase (GGT), Red Blood Cell Count (RBC), Hematocrit (HCT), Mean Cell Volume (MCV), Mean Cell Hemoglobin (MCH), Mean Cell Hemoglobin Concentration (MCHC), Red Cell Distribution Width (RDW), Platelets, Mean Platelet Volume (MPV), Monocytes, Neutrophils, Lymphocytes, Eosinophils, Basophils, Hemoglobin, Ferritin, Total Iron Binding Capacity (TIBC), Iron, Transferrin Saturation (TS), Folate, Vitamin B12, Calcium, Vitamin D, Magnesium, Red Blood Cell Magnesium, Potassium, Sodium, Creatine Kinase (CK), Testosterone, Free Testosterone, Dehydroepiandrosterone-sulfate (DHEAS), Cortisol, Sex Hormone Binding Globulin (SHBG), Albumin, Glucose, Total Cholesterol, High-Density Lipoprotein cholesterol (HDL), Low-Density Lipoprotein cholesterol (LDL), Triglycerides, White Blood Cell Count (WBC), High Sensitivity C-Reactive Protein (hsCRP). Secretory Immunoglobulin A (sIgA) was measured in saliva collected from participants.

ELIGIBILITY:
Inclusion Criteria:

1. Employees and family and friends of employees.
2. Adults committed to attend all of the sessions and follow the instructions described in Experimental Design.
3. Participants of both genders and of ages >18 will be included.
4. Participants with the best chance to benefit from taking the product, i.e., participants that are not in the optimal health/level as per answers in the health questionnaire, but that are not diseased.

Exclusion Criteria

1. Pregnant and nursing women.
2. Those currently taking 4Life TF Plus and/or other supplements containing vitamins, minerals, and essential fatty acids (EPA/DHA, fish oil, omega 3), and those that have taken any of these supplements up to 1 month prior to first study visit.
3. Those participants that reported to take daily medications to treat a chronic condition. However, birth control pill does not count.
4. Those participants with allergies to any of the ingredients of the product including high sensitivity to lactose.
5. Participants that smoke and with body mass index (BMI) either < 19 or > 30 will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Salivary IgA | 12 weeks
  Secretory Immunoglobulin A (sIgA) was measured in saliva collected from participants.
Serum folate level | 12 weeks
  Serum folate level was measured in blood sample collected from participants
Serum vitamin B12 level | 12 weeks
  Serum vitamin B12 level was measured in blood sample collected from participants
Serum vitamin D level | 12 weeks
  Serum vitamin D level was measured in blood sample collected from participants

SECONDARY OUTCOMES:
Alanine Aminotransferase (ALT) Activity | 12 weeks
  ALT activity is measured in blood sample collected from participants. ALT, AST, and GGT are important biomarkers for liver function and commonly used for safety assessment
Aspartate Aminotransferase (AST) activity | 12 weeks
  AST activity is measured in blood sample collected from participants. ALT, AST, and GGT are important biomarkers for liver function and commonly used for safety assessment
Gamma-Glutamyl Transpeptidase (GGT) activity | 12 weeks
  GGT activity is measured in blood sample collected from participants. ALT, AST, and GGT are important biomarkers for liver function and commonly used for safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: David Vollmer, PhD, Study Chair — 4Life Research, LLC
Locations (1):
- 4Life Research, Sandy City, Utah, United States

IPD SHARING:
Plan to Share IPD: No